CLINICAL TRIAL: NCT04799938
Title: Effect of Exercise on GDF-15 Levels in Prediabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACTİVE GD-15
Record Dates: First submitted 2021-03-07; First posted 2021-03-16 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: PreDiabetes
Keywords: GDF-15; Physical Exercise; Prediabetes
MeSH Terms: conditions — Prediabetic State; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Exercise intervention will be applied to intervention group All participiants will be applied to standard recommendations
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- İntevention group (Active Comparator): Prediabetic patients with age 30-50 and overweight Standart recommendations Exercise intervention will be made.
  Interventions: Behavioral: Exercise
- Control group (No Intervention): Prediabetic patients with age 30-50 and overweight Only Standart recommendations
- Metformin Group (No Intervention): Prediabetic patients who received metformin Standart recommendations

INTERVENTIONS:
Behavioral: Exercise — 180 minutes of moderate-intensity exercise per week
  Arms: İntevention group

SUMMARY:
The aim of this study is to evaluate whether there is a change in GDF-15 levels in individuals with prediabetes at the 2nd hour after the first exercise and after a 12-week exercise program with guide-based exercise programs.

DETAILED DESCRIPTION:
GDF-15, which has anorexigenic effects, increases with exercise. In prediabetic patients, GDF-15 is higher than healthy controls. The effect of exercise on GDF-15 levels in prediabetic patients is unknown.

The aim of this study is to evaluate whether there is a change in GDF-15 levels after the application of guideline-based exercise programs in individuals with prediabetes at the 2nd hour after the first exercise and after a 12-week exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 30-34.9 kg / m2
* Sedentary life-style (Physical activity below 300 kcal / day will be assessed by Minnesota Leisure Physical Activity Questionnaire)
* Those who have sufficient motivation to participate in the exercise program (will be evaluated by face-to-face interview by the researchers)
* Having the same weight for 6 months before participating in the study (± 2.5 kg)
* Those diagnosed with prediabetes by oral glucose tolerance test and / or HbA1c measurement will be included.

Exclusion Criteria:

* Serious medical condition (e.g. advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.)
* Having cardiovascular disease
* Having diabetes
* Using metformin
* Taking hormone replacement therapy
* less than 1 year life expectancy
* HIV positivity
* Substance use
* Functional dependence
* Cognitive weakness
* Those with other diseases that will affect the study result (respiratory diseases, muscle diseases, etc.)
* Those who use drugs or supplements that will affect the results of the study

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Level of Growth Diferantiation Factor-15 | 12 weeks
  Level of Growth Diferantiation Factor-15

SECONDARY OUTCOMES:
Level of VO2max | 12 weeks
  Level of VO2max

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Han Training and Rsearch Hospital
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Turkey (Türkiye)